CLINICAL TRIAL: NCT07173231
Title: Comparisons Between Virtual Reality and Hypno-Virtual Reality for Procedural Pain and Anxiety During a Diagnostic Hysteroscopy: A Pilot Randomized Controlled Trial
Brief Title: Use of VR for Diagnostic Hysteroscopy
Acronym: VR-HYSTERO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Le May, Principal investigator, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VR-HYSTERO
Record Dates: First submitted 2025-08-27; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hysteroscopy; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This pilot RCT study is mainly designed to test the feasibility and acceptability of the intervention, design and procedures. Therefore, we did not calculate a specific sample size to detect statistically significant differences. Instead, a convenience sample of 45 participants (15 per group) was selected based on established recommendations for pilot studies, which suggest that 12 participants per arm is adequate to evaluate feasibility and provide preliminary results for planning a future clinical trial (Julious, 2005). The sample size was also determined based on practical considerations related to the recruitment capacity and the study resources, as each group will include approximately 15 participants, representing about 30% of the 150 diagnostic hysteroscopy procedures performed annually at the CHU Sainte-Justine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersive Virtual Reality Distraction (IVR) (Experimental): Use of IVR during diagnostic hysteroscopy
  Interventions: Device: Immersive Virtual Reality Distraction (IVR)
- Hypno-Virtual Reality distraction (HVR) (Experimental): Use of HVR during diagnostic hysteroscopy
  Interventions: Device: Hypno-Virtual Reality Distraction (HVR)
- Usual Care Treatment (Active Comparator): Standard protocol offered at CHU Ste-Justine's Hospital before a diagnostic hysteroscopy procedure
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Device: Immersive Virtual Reality Distraction (IVR) — The first experimental group will receive the INSPIRE® IVR intervention in addition to usual care. Developed by Paperplane Therapeutics®, INSPIRE® is specifically designed to help manage pain and anxiety in clinical settings. This intervention integrates immersive virtual environments with sensor-guided deep breathing techniques to engage the parasympathetic nervous system and promote relaxation. Within a calming forest environment, participants are guided to synchronize their breathing with the movement of a feather, encouraging breath control and relaxation. The immersive experience is enhanced through personalized therapeutic content and calming visual and auditory stimuli, helping to reduce anxiety while minimizing the risk of cybersickness. This program has been endorsed by a multidisciplinary team of healthcare professionals.
  Arms: Immersive Virtual Reality Distraction (IVR)
Device: Hypno-Virtual Reality Distraction (HVR) — The second experimental group will receive the HVR intervention in addition to usual care. This intervention, developed by HypnoVR, consists of a VR visual scenario combined with hypnotic verbal guidance specifically designed to reduce pain and anxiety during medical procedures. It is delivered through a validated and clinically approved HVR headset. The intervention includes reassuring and calming verbal suggestions aimed at helping participants regulate their emotions and manage anxiety throughout the procedure. Participants will be able to choose from 11 different visual scenarios, select their preferred language, and choose between a male or female voice for the hypnotic guidance. 6 different musical soundtracks will also be available to personalize the experience more.
  Arms: Hypno-Virtual Reality distraction (HVR)
Other: Usual Care Group — The usual care group will only receive the standard preparation, which includes pre-treatment with Tylenol (1000mg) , Naproxen (500mg) and Ativan (1 mg) administered one hour prior to the procedure.
  Arms: Usual Care Treatment

SUMMARY:
Background: Hysteroscopy (HSC) is a minimally invasive gynecological procedure that is considered to be the gold standard for diagnosing and treating intrauterine pathologies. In recent years, its use in outpatient settings for diagnosis has grown significantly due to its efficiency, low complication rate, and good patient acceptability. However, many patients still report significant pain and anxiety during the procedure. Despite advances in instrumentation and technique, pain remains a key reason for procedural failure, often worsened by preprocedural anxiety. While pharmacological strategies can be used to address this issue, they are not always suitable due to lack of effectiveness or feasibility. As a result, non-pharmacological approaches such as virtual reality (VR) and hypnosis are being increasingly explored. VR has shown potential in reducing pain and anxiety during medical procedures, and its combination with hypnosis may offer enhanced benefits, though current evidence is limited.

Objective: This pilot study aims to assess the effectiveness of immersive virtual reality (IVR) and Hypno-VR (HVR) in managing pain and anxiety during diagnostic HSC and to evaluate the feasibility and acceptability of both IVR and HVR interventions in an outpatient clinical setting.

Methods: This pilot randomized controlled trial (RCT) will follow a three-arm parallel design to compare: 1- standard care, 2- IVR + standard care, and 3- HVR + standard care, during diagnostic HSC. A total of 45 participants (15/arm) will be recruited from the CHU Sainte-Justine's gynecology clinic and randomly assigned to one of the three groups. Primary outcomes will concern feasibility and acceptability including satisfaction of both patients and healthcare professionals. Secondary outcomes will assess self-reported pain and anxiety, physiological responses, procedure duration, procedure failure, and conversion rate from the "no-touch" vaginoscopy technique to traditional tools like the speculum and tenaculum. Demographic characteristics will also be explored as potential moderators of intervention effectiveness.

Results/Conclusion: This pilot study will provide preliminary data on the effects of IVR and HVR on procedural pain and anxiety during diagnostic HSC. It will also assess the feasibility and the acceptability of integrating these interventions into an outpatient setting. The findings will provide essential data in preparation for a larger clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years old
* Speak and read French or English
* Scheduled to undergo a diagnostic hysteroscopy

Exclusion Criteria:

* Having a diagnosis of epilepsy
* Recent ophthalmologic surgery (< 1month) or any ophtalmologic problems that could interfere with the patient's ability to use the VR technology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Completion rate of the planned intervention | To be reported at the end of the intervention, about 2 minutes after the end of the hysteroscopy procedure (T2)
  Completion rate of the planned intervention will be assessed as the proportion of participants who complete their allocated intervention out of the total number of participants randomized.
Recruitment rate | To be reported right before the procedure, at baseline (T0)
  Recruitment rate will be assessed as the proportion of patients who consent to participate out of the total number of HSC procedures performed.
The healthcare professionals' satisfaction level | To be reported at the end of the intervention, about 2 minutes after the end of the hysteroscopy procedure (T2)
  The healthcare professionals' satisfaction level will be assessed using a customized questionnaire comprising 7-10 items, depending on the intervention used. Each item will be rated on a four-point Likert scale, ranging from "Strongly agree" to "Strongly disagree," evaluating their satisfaction with the intervention and its perceived impact on the procedure (T2).
The patient's satisfaction level | To be reported at the end of the intervention, about 2 minutes after the end of the hysteroscopy procedure (T2)
  The patient's satisfaction level towards the intervention will be assessed using a Verbal Numerical Rating Scale (VNRS), ranging from 0 to 10, where 0 indicates "very dissatisfied" and 10 indicates "very satisfied." Patients will be asked the following question: "Considering anxiety relief, pain relief, side effects, and emotional recovery, how satisfied were you with the treatments you received during the procedure?" (T2).
Patient's acceptability towards the intervention | To be reported at the end of the intervention, about 2 minutes after the end of the hysteroscopy procedure (T2)
  The patient's acceptability towards the intervention will be assessed using the Treatment Acceptability & Preference (TAP) questionnaire: 10 questions (6 Likert-scale items from 0 to 4 and 4 open-ended questions). These questions focus on acceptability, satisfaction, ease of use, perceptions, and suggestions for improvement (T2).

SECONDARY OUTCOMES:
Pain intensity | Assessments will be conducted at baseline (T0), 2 minutes after the intervention (T2), and one week post-intervention (T3). The T3 assessment will be performed by a research assistant.
  Pain intensity will be measured using the Verbal Numerical Rating Scale (VNRS), a self-report scale ranging from 0 to 10, where 0 represents no pain and 10 corresponds to the worst pain imaginable.
Anxiety intensity | Measurements will be taken at baseline (T0), 2 minutes after the intervention (T2), and one week later (T3). The T3 evaluation will be conducted by a research assistant through the participant's preferred mode of communication.
  Anxiety intensity will be assessed using a validated self-report scale (VNRS) ranging from 0 to 10, where 0 signifies no anxiety and 10 indicates the highest possible level of anxiety.
Change in heart rate | Heart rate will be measured right before the procedure, at baseline (T0) and about 2 minutes after the end of the hysteroscopy procedure (T2).
  Change in heart rate will be measured by using COVIDIEN Nellcor pulse oxygen saturation meter, an approved and validated device (T0, T2).
Failure of hysteroscopy | To be reported during the procedure (T1)
  Failure of hysteroscopy will be assessed by recording the number of procedures that are not completed as intended or that require rescheduling.
Required time for the procedure | To be reported during the procedure (T1)
  Required time for the procedure will be measured in minutes, starting from the insertion of the hysteroscope intravaginally to its removal, and will be recorded by the research nurse.
Demographic and clinical characteristics | Demographic and clinical characteristics will be assessed at baseline (T0)
  Demographic and clinical characteristics associated with greater benefit from the experimental interventions will be assessed by analyzing variables such as age, menopausal status, previous gynecological history, and prior experience with VR or hypnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May PhD, Principal Investigator — St. Justine's Hospital

REFERENCES:
- [Background] Rousseaux F, Bicego A, Ledoux D, Massion P, Nyssen AS, Faymonville ME, Laureys S, Vanhaudenhuyse A. Hypnosis Associated with 3D Immersive Virtual Reality Technology in the Management of Pain: A Review of the Literature. J Pain Res. 2020 May 21;13:1129-1138. doi: 10.2147/JPR.S231737. eCollection 2020. PMID 32547176
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Babbar S, Oyarzabal AJ. The Application of Hypnosis in Obstetrics. Clin Obstet Gynecol. 2021 Sep 1;64(3):635-647. doi: 10.1097/GRF.0000000000000635. PMID 34323237
- [Background] Cohen N, Nasra LA, Paz M, Kaufman Y, Lavie O, Zilberlicht A. Pain and anxiety management with virtual reality for office hysteroscopy: systemic review and meta-analysis. Arch Gynecol Obstet. 2024 Apr;309(4):1127-1134. doi: 10.1007/s00404-023-07261-9. Epub 2023 Nov 2. PMID 37917158
- [Background] Sewell T, Fung Y, Al-Kufaishi A, Clifford K, Quinn S. Does virtual reality technology reduce pain and anxiety during outpatient hysteroscopy? A randomised controlled trial. BJOG. 2023 Nov;130(12):1466-1472. doi: 10.1111/1471-0528.17550. Epub 2023 May 23. PMID 37218438
- [Background] Baradwan S, Alshahrani MS, AlSghan R, Alyafi M, Elsayed RE, Abdel-Hakam FA, Moustafa AA, Hussien AE, Yahia OS, Shama AA, Magdy AA, Abdelhakim AM, Badran H. The effect of virtual reality on pain and anxiety management during outpatient hysteroscopy: a systematic review and meta-analysis of randomized controlled trials. Arch Gynecol Obstet. 2024 Apr;309(4):1267-1280. doi: 10.1007/s00404-023-07319-8. Epub 2024 Jan 2. PMID 38165441
- [Background] Deo N, Khan KS, Mak J, Allotey J, Gonzalez Carreras FJ, Fusari G, Benn J. Virtual reality for acute pain in outpatient hysteroscopy: a randomised controlled trial. BJOG. 2021 Jan;128(1):87-95. doi: 10.1111/1471-0528.16377. Epub 2020 Jul 22. PMID 32575151
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Tas FQ, van Eijk CAM, Staals LM, Legerstee JS, Dierckx B. Virtual reality in pediatrics, effects on pain and anxiety: A systematic review and meta-analysis update. Paediatr Anaesth. 2022 Dec;32(12):1292-1304. doi: 10.1111/pan.14546. Epub 2022 Sep 1. PMID 35993398
- [Background] Paulo AAS, Solheiro MHR, Paulo COS, Afreixo VMA. What proportion of women refers moderate to severe pain during office hysteroscopy with a mini-hysteroscope? A systematic review and meta-analysis. Arch Gynecol Obstet. 2016 Jan;293(1):37-46. doi: 10.1007/s00404-015-3836-5. Epub 2015 Aug 8. PMID 26253336
- [Background] Samy A, Nabil H, Abdelhakim AM, Mahy ME, Abdel-Latif AA, Metwally AA. Pain management during diagnostic office hysteroscopy in postmenopausal women: a randomized study. Climacteric. 2020 Aug;23(4):397-403. doi: 10.1080/13697137.2020.1742685. Epub 2020 Apr 17. PMID 32299254
- [Background] Riemma G, Schiattarella A, Colacurci N, Vitale SG, Cianci S, Cianci A, De Franciscis P. Pharmacological and non-pharmacological pain relief for office hysteroscopy: an up-to-date review. Climacteric. 2020 Aug;23(4):376-383. doi: 10.1080/13697137.2020.1754388. Epub 2020 May 12. PMID 32396751
- [Background] Ghamry NK, Samy A, Abdelhakim AM, Elgebaly A, Ibrahim S, Ahmed AA, Abdelbaky WH, Abdallah KM, Badawy MA, Mohammed AH, Hamza M. Evaluation and ranking of different interventions for pain relief during outpatient hysteroscopy: A systematic review and network meta-analysis. J Obstet Gynaecol Res. 2020 Jun;46(6):807-827. doi: 10.1111/jog.14221. Epub 2020 Feb 23. PMID 32088931
- [Background] Bracken O, Woodsmith A, Newell M. Pharmacological and non-pharmacological interventions for pain control in outpatient hysteroscopy: A systematic review. Eur J Obstet Gynecol Reprod Biol. 2025 Mar;306:35-46. doi: 10.1016/j.ejogrb.2025.01.004. Epub 2025 Jan 5. PMID 39787964
- [Background] Carta G, Palermo P, Marinangeli F, Piroli A, Necozione S, De Lellis V, Patacchiola F. Waiting time and pain during office hysteroscopy. J Minim Invasive Gynecol. 2012 May-Jun;19(3):360-4. doi: 10.1016/j.jmig.2012.01.017. Epub 2012 Mar 3. PMID 22387163
- [Background] Law, J.Y.P. (2023). Pain relief in hysteroscopy. Hong Kong Journal of Gynaecology, Obstetrics and Midwifery, 23(1). DOI: https://doi.org/10.12809/hkjgom.23.1.08
- [Background] Vitale SG, Alonso Pacheco L, Haimovich S, Riemma G, De Angelis MC, Carugno J, Lasmar RB, Di Spiezio Sardo A. Pain management for in-office hysteroscopy. A practical decalogue for the operator. J Gynecol Obstet Hum Reprod. 2021 Jan;50(1):101976. doi: 10.1016/j.jogoh.2020.101976. Epub 2020 Nov 6. PMID 33166706
- [Background] Vitale SG, Caruso S, Ciebiera M, Torok P, Tesarik J, Vilos GA, Cholkeri-Singh A, Gulino FA, Kamath MS, Cianci A. Management of anxiety and pain perception in women undergoing office hysteroscopy: a systematic review. Arch Gynecol Obstet. 2020 Apr;301(4):885-894. doi: 10.1007/s00404-020-05460-2. Epub 2020 Mar 5. PMID 32140807
- [Background] de Campos BF, Benetti-Pinto CL, Yela DA. Nurse support for pain and anxiety control in women undergoing diagnostic hysteroscopy: a randomized clinical trial. Menopause. 2023 Sep 1;30(9):927-932. doi: 10.1097/GME.0000000000002226. Epub 2023 Jul 25. PMID 37490654
- [Background] Estadella Tarriel J, Perello Capo J, Simo Gonzalez M, Bailon Queiruga M, Real Gatius J, Gomis-Pastor M, Marre D, Llurba Olive E. Effectiveness of Virtual Reality in Reducing Pain and Stress During Office Hysteroscopy: A Randomized Controlled Trial. Healthcare (Basel). 2025 Jan 12;13(2):131. doi: 10.3390/healthcare13020131. PMID 39857158
- [Background] Cicinelli E. Hysteroscopy without anesthesia: review of recent literature. J Minim Invasive Gynecol. 2010 Nov-Dec;17(6):703-8. doi: 10.1016/j.jmig.2010.07.003. PMID 20955981
- [Background] Coimbra AC, Falcao V, Pinto P, Cavaco-Gomes J, Fernandes AS, Martinho M. Predictive Factors of Tolerance in Office Hysteroscopy - a 3-Year Analysis from a Tertiary Center. Rev Bras Ginecol Obstet. 2023 Jan;45(1):38-42. doi: 10.1055/s-0043-1764361. Epub 2023 Mar 6. PMID 36878251
- [Background] Amer-Cuenca JJ, Marin-Buck A, Vitale SG, La Rosa VL, Caruso S, Cianci A, Lison JF. Non-pharmacological pain control in outpatient hysteroscopies. Minim Invasive Ther Allied Technol. 2020 Feb;29(1):10-19. doi: 10.1080/13645706.2019.1576054. Epub 2019 Feb 22. PMID 30794005
- [Background] Ignaszak-Kaus, N., Chmaj-Wierzchowska, K., Nowak, A., Wszolek, K., and Wilczak, M. (2022). An Overview of Outpatient Hysteroscopy. Clinical and Experimental Obstetrics & Gynecology, 49(8), 181. https://doi.org/10.31083/j.ceog4908181.
- [Background] Guraslan H, Senturk MB, Dogan K, Yuksel B, Kaya C, Karacan T, Karabay Akgul O, Ceylan Y. Diagnostic office hysteroscopy; why is it still painful procedure despite the surgical experience and mini-hysteroscope? J Obstet Gynaecol Res. 2022 Jun;48(6):1418-1425. doi: 10.1111/jog.15219. Epub 2022 Mar 10. PMID 35274418
- [Background] Buzzaccarini G, Alonso Pacheco L, Vitagliano A, Haimovich S, Chiantera V, Torok P, Vitale SG, Lagana AS, Carugno J. Pain Management during Office Hysteroscopy: An Evidence-Based Approach. Medicina (Kaunas). 2022 Aug 20;58(8):1132. doi: 10.3390/medicina58081132. PMID 36013599
- [Background] Bakour SH, Jones SE, O'Donovan P. Ambulatory hysteroscopy: evidence-based guide to diagnosis and therapy. Best Pract Res Clin Obstet Gynaecol. 2006 Dec;20(6):953-75. doi: 10.1016/j.bpobgyn.2006.06.004. Epub 2006 Nov 20. PMID 17116420
- [Background] Orlando MS, Bradley LD. Implementation of Office Hysteroscopy for the Evaluation and Treatment of Intrauterine Pathology. Obstet Gynecol. 2022 Sep 1;140(3):499-513. doi: 10.1097/AOG.0000000000004898. Epub 2022 Aug 3. PMID 35926213